CLINICAL TRIAL: NCT00984347
Title: Breast Pump Nipple Stimulation Versus Pitocin for Induction of Labor: Efficacy, Safety and Satisfaction
Brief Title: Breast Stimulation Versus Pitocin for Induction of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Sciaky-Tamir Yael, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280808-HMO-CTIL
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Labor Induction
Keywords: nipple stimulation; Oxytocin; induction of labor; term pregnancies; grandmultipara; VBAC; PROM; comparison of two methods for induction of labor
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin induction (Active Comparator): women in need for induction of labor due to medical indications, will receive continuous IV oxytocin
  Interventions: Drug: Oxytocin
- Breast Stimultion (Active Comparator): nipple stimulation with a breast pump, calibrated at the lowest suction strength,operated alternately: 15 min one breast, 15 min second breast, 15 min rest, till appearance of regular uterine contractions (3 contractions in 10 min). the manipulation will continue for 3 hours of regular contractions.
  Interventions: Procedure: breast pump nipple stimulation

INTERVENTIONS:
Drug: Oxytocin — For low risk group (women at deliveries 1-5):
  IV oxytocin 10IU/1000ml standard sol. starting at 2MU/MIN and augmenting 2MU every 20 min.
  For high risk group (grandmultiparas [6th delivery and up] or women with a previous cesarean section)
  IV oxytocin 5IU/1000ml standard sol. starting at 1MU/MIN augmenting 1MU every 20 MIN - in accordance with the department's protocol
  Other Names: Oxytocin for injection 10u/ml Rotex Medica
  Arms: Oxytocin induction
Procedure: breast pump nipple stimulation — breast pump calibrated at lowest suction strength, operated alternately: 15 min one breast, 15 min second breast, 15 min rest
  Arms: Breast Stimultion

SUMMARY:
The purpose of the trial is to compare nipple stimulation with a breast pump to pitocin for induction of labor in term pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* completed 37 weeks gestation
* singleton pregnancy
* reassuring fetal heart rate at admission monitor

Exclusion Criteria:

* multiple pregnancies
* known fetal malformations
* non reassuring NST
* polyhydramnios (AFI>220)
* oligohydramnios
* PET
* IUGR
* macrosomia (EFW >4000g)
* antepartum bleeding
* maternal fever

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
time from induction to delivery | 24h

SECONDARY OUTCOMES:
fetal distress (monitor assessment, cord ph) | 24 h
cesarean section rate | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Drorith Hochner-Celnikeir, MD, Study Chair — Hadasah Medical Organization
Locations (1):
- Hadassah University Hospital Mt. Scopus, Jerusalem, Israel